CLINICAL TRIAL: NCT00696488
Title: Measuring Adherence To Topical 5-Fluorouracil in a Clinic Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000156; 31358
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluorouracil 0.5% (Experimental): each subject will receive the study medication: Carac® 0.5% Fluorouracil, a standard treatment for actinic keratoses. Carac® will be dispensed to the subjects in the original tube with MEMS electronic monitoring caps attached. Subjects will be asked to apply the medication daily to AK lesions
  Interventions: Drug: Fluorouracil 0.5%

INTERVENTIONS:
Drug: Fluorouracil 0.5% — Subjects will apply the smallest amount of study medication possible that is just sufficient to cover all of the affected areas daily to AK lesions
  Other Names: Carac

SUMMARY:
The purpose of this research study is to measure adherence to the study drug (Carac) for the treatment of actinic keratoses.

DETAILED DESCRIPTION:
The purpose of this research study is to measure adherence to the study drug for the treatment of actinic keratoses. The study drug is 5-Fluorouracil (Carac®); it will be used in this study to treat actinic keratoses on the face and anterior scalp. This proposed study will evaluate adherence to topical Carac® in 20 adults age 50 or greater with actinic keratoses from a clinic population. Adherence data will be collected by the MEMS cap (Medication Event Monitoring System

ELIGIBILITY:
Inclusion Criteria:

* Any male or female 50 years of age or older with moderate to severe actinic keratoses of the face and anterior scalp diagnosed by a dermatologist will be eligible for participation.

Exclusion Criteria:

* Age less than 50.
* Known allergy or sensitivity to topical Carac® in the subject.
* Inability to complete all study-related visits.
* Introduction of any other prescription medication, topical or systemic, for actinic keratosis while participating in the study.
* Subjects should not receive surgical or cryotherapy while participating in the study.
* Pregnant women, women who are breast feeding, or women of child bearing potential who are not practicing two acceptable methods of birth control

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-04; Primary Completion 2007-08 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yentzer B, Hick J, Williams L, Inabinet R, Wilson R, Camacho FT, Russell GB, Feldman SR. Adherence to a topical regimen of 5-fluorouracil, 0.5%, cream for the treatment of actinic keratoses. Arch Dermatol. 2009 Feb;145(2):203-5. doi: 10.1001/archdermatol.2008.562. No abstract available. PMID 19221274

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluorouracil 0.5%
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fluorouracil 0.5%
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 67 [51 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Carac® in Subjects With Moderate to Severe Actinic Keratosis.
Description: Measure of adherence by MEMS caps and the % of total prescribed doses that were actually used
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: percentage of prescribed doses
Arm/Group | Fluorouracil 0.5%
Number analyzed (Participants) | 20
percentage of prescribed doses | 86 [54 to 100]

ADVERSE EVENTS:
Arm/Group | Fluorouracil 0.5%
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluorouracil 0.5% (N=20)
Burning of skin (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes